CLINICAL TRIAL: NCT00134082
Title: Pilot Study of Rituximab, High Dose Cyclophosphamide, and GM-CSF Based Immunotherapy for Relapsed Hodgkin's Lymphoma
Brief Title: Rituximab and Cyclophosphamide Followed by Vaccine Therapy in Treating Patients With Relapsed Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0528; P50CA096888 (NIH); P30CA006973 (NIH); NA_00035358 (Other: JHMIRB)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Cyclophosphamide

ARMS (1):
- Immunotherapy (Experimental): All participants received two days of rituximab, then four days of high-dose cyclophosphamide followed by filgrastim. Participants then received six doses of KGEL vaccine over 24 weeks interspersed with four additional doses of rituximab.
  Interventions: Biological: KGEL vaccine; Biological: Filgrastim; Biological: Rituximab; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: KGEL vaccine — Vaccine was administered at weeks 0, 4, 8, 12, 16, and 24 at a dose of 1 x 10^8 cells per dose. The first dose was given on Day +1.
Biological: Filgrastim — 5 mcg/kg/day starting on Day +6 until ANC is >= 1000/mcL.
  Other Names: G-CSF
Biological: Rituximab — 375 mg/m^2/day on Days -10, -7, and at weeks 4, 5, 6, and 7.
  Other Names: Rituxan
Drug: Cyclophosphamide — 50 mg/kg/day on Day -3, -2, -1, and 0.
  Other Names: Cytoxan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells either by killing the cells or by stopping them from dividing. Vaccines made from another person's cancer cells may help the body build an effective immune response to kill cancer cells. Giving rituximab together with chemotherapy and vaccine therapy may kill more cancer cells

PURPOSE: This phase I/II trial is studying how well giving rituximab together with cyclophosphamide and vaccine therapy works in treating patients with relapsed Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of rituximab and high-dose cyclophosphamide followed by vaccine therapy comprising an allogeneic vaccine that expresses Hodgkin's tumor antigens and sargramostim (GM-CSF) (KGEL vaccine) as salvage therapy in patients with relapsed Hodgkin lymphoma.
* Determine the immunologic response to this vaccine in these patients.

Secondary

* Determine the 3-year relapse-free and overall survival of patients treated with this regimen.
* Determine the patterns of cellular immune reconstitution in patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive rituximab IV on days -10 and -7 and then on days 29, 36, 43, and 50 (weeks 4-7) and high-dose (transplant-dose) cyclophosphamide IV on days -3 to 0 without stem cell rescue. Patients receive filgrastim (G-CSF) subcutaneously once daily beginning on day 6 and continuing until blood counts recover. Patients also receive vaccine therapy comprising an allogeneic vaccine that expresses Hodgkin's tumor antigens and sargramostim (GM-CSF) (KGEL vaccine) intradermally on day 1, and weeks 4, 8, 12, 16, and 24.

After completion of high-dose cyclophosphamide, patients are followed every 3 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classical Hodgkin's lymphoma
* Relapsed disease with achievement of at least a partial response or a metabolic response to most recent salvage therapy

  * No primary induction failure, defined as disease progression during or within 2 months after completion of first-line therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL* NOTE: *Unless due to lymphoma or Gilbert's syndrome

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* Ejection fraction ≥ 45% by echocardiogram or MUGA

Pulmonary

* DLCO ≥ 50% of predicted (corrected for alveolar volume)

Immunologic

* No known HIV positivity
* No active infection requiring oral or IV antibiotics
* No autoimmune or other disease requiring long-term systemic steroids or other long-term immunosuppressants

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to tolerate high-dose therapy
* No other malignancy within the past 3 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior bone marrow transplantation

Endocrine therapy

* Not specified

Radiotherapy

* Concurrent radiotherapy for disease progression after high-dose cyclophosphamide allowed at the discretion of the principal investigator

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ambinder, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was a screen failure.
Period: Overall Study
Arm/Group | Immunotherapy
Started | 30
Completed | 27
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Immunotherapy
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 39.5 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3-5 Adverse Events
Description: Number of participants who experienced at least one grade 3-5 adverse event by CTCAE 3.0 that was attributed to protocol intervention.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immunotherapy
Number analyzed (Participants) | 30
Participants | 6

2. Primary Outcome: Percentage of Participants With an Increase in Frequency of LMP2-specific CD8+ T Cells
Description: Percentage of participants with an increase in frequency of LMP2-specific CD8+ T cells. Increase in frequency is defined as at least one order of magnitude higher than baseline measurement.
Time Frame: Change from 3 months to 6 months
Population: Although the specimens were collected per protocol, they were not interpretable and therefore no data was collected to assess this outcome measure
Arm/Group | Immunotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival
Description: Median number of months that participants were alive (overall survival) and alive without disease relapse or new diagnosis of myelodysplasia or acute leukemia (event-free survival).
Time Frame: Up to 6 years
Measure: Median (Full Range); unit: months
Arm/Group | Immunotherapy
Number analyzed (Participants) | 30
months
  Overall survival | 31.5 [12.2 to 70.9]
  Event-free survival | 24.1 [4.9 to 63]

4. Secondary Outcome: Days to Neutrophil and Platelet Engraftment
Description: Median number of days to absolute neutrophil count (ANC) >= 500/mcL and platelet count >=20000/mcL.
Time Frame: Up to 46 days
Measure: Median (Full Range); unit: days
Arm/Group | Immunotherapy
Number analyzed (Participants) | 30
days
  Days until ANC >= 500mcL | 17 [10 to 26]
  Days until Platelet Count >=20000/mcL | 21.5 [10 to 46]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: The following adverse events only were collected on this study:
  * All adverse events attributed to the vaccine
  * All grade 3-5 nonhematologic toxicities until 30 days post last dose of vaccine
  * Any hospitalization or death until 30 days post last dose of vaccine
  * Grade 3-4 neutropenia until 1 year post completion of high-dose cyclophosphamide
Arm/Group | Immunotherapy
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy (N=30)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Influenza A (Infections and infestations) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 9 (9)
Cytopenia (Investigations) | 1 (1)
Rigors (General disorders) | 1 (1)
Pain - back (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombus (Vascular disorders) | 1 (1)
Infection, not specified (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy (N=30)
Anemia (Investigations) | 2 (28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Bruising (Skin and subcutaneous tissue disorders) | 2 (3)
Dizziness (Nervous system disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Fatigue (General disorders) | 21 (26)
Fever (General disorders) | 3 (4)
Headache (General disorders) | 12 (28)
Injection site reaction (Skin and subcutaneous tissue disorders) | 30 (258)
Leukopenia (Investigations) | 2 (16)
Lymphopenia (Investigations) | 4 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutropenia (Investigations) | 29 (110)
Pain - knee (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - thigh (Musculoskeletal and connective tissue disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (8)
Thrombocytopenia (Investigations) | 4 (31)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weakness (Nervous system disorders) | 3 (3)
Xerosis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes